CLINICAL TRIAL: NCT03022916
Title: Real-World Evaluation of the Effect of Jublia on Nail Polish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Boni Elewski, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: X150817005
Record Dates: First submitted 2015-10-16; First posted 2017-01-18 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Evaluation of Jublia on Nail Polish With Healthy Toenails
Keywords: toenail polish; jublia
MeSH Terms: interventions — efinaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nail Polish + Efinaconazole Solution (Active Comparator): One big toe will receive application of Efinaconazole Solution on top of nail polish (without the presence of a top coat or base coat)
  Interventions: Drug: Nail Polish + Efinaconazole Solution
- Nail Polish Only (Placebo Comparator): Both big toes will use nail polish only
  Interventions: Other: Nail polish
- Base Coat + Nail Polish + Top Coat + Efinaconazole Solution (Active Comparator): One big toe will receive application of Efinaconazole solution on top of nail polish with base coat and top coat.
  Interventions: Drug: Base Coat + Nail Polish + Top Coat + Efinaconazole Solution
- Nail Polish + Top Coat + Efinaconazole Solution (Active Comparator): One big toe will receive application of Efinaconazole solution on top of nail polish with top coat.
  Interventions: Drug: Nail Polish + Top Coat + Efinaconazole Solution

INTERVENTIONS:
Drug: Nail Polish + Efinaconazole Solution — Application of Jublia to the nail of one big toe on top of the nail polish
  Other Names: Jublia
  Arms: Nail Polish + Efinaconazole Solution
Other: Nail polish — Application of nail polish only to both big toe nails
  Arms: Nail Polish Only
Drug: Base Coat + Nail Polish + Top Coat + Efinaconazole Solution — Application of Jublia to the nail of one big toe on top of the nail polish with layers of top coat and base coat
  Other Names: Jublia
  Arms: Base Coat + Nail Polish + Top Coat + Efinaconazole Solution
Drug: Nail Polish + Top Coat + Efinaconazole Solution — Application of Jublia to the nail of one big toe on top of the nail polish with layer of top coat
  Other Names: Jublia
  Arms: Nail Polish + Top Coat + Efinaconazole Solution

SUMMARY:
A recent publication using cadaver nails suggests that Jublia application has a negative effect on nail polish texture.

DETAILED DESCRIPTION:
It is believed that investigating the affect of Jublia is an important question with regards to how it affects how various nail polished and top coats will be used.

ELIGIBILITY:
Inclusion Criteria:

* Exhibit distal lateral subungual onychomycosis (DLSO)
* Has the informed consent been signed and patient's questions answered.
* Age ≥ 18
* Patient willing and able to participate for the full duration of the study
* No onychomycosis
* Greater than 4 weeks from prior major surgery for any indication
* Willing to abstain from:
* The application of other topical medications or cosmetic products to the toenail
* Professional pedicures for the duration of the study.
* Females of childbearing potential must:
* Have been using adequate contraception (abstinence, IUD, birth control pills or spermicidal gel with diaphragm or condom) since their last menses
* Agree to continue using adequate means of contraception (abstinence, IUD, birth control pills or spermicidal gel with diaphragm or condom) for the duration of study participation
* Females are not considered to be of childbearing potential if they are at least 1 year postmenopausal or have had a tubal ligation, bilateral oophorectomy or hysterectomy.

Exclusion Criteria:

* Active onychomycosis of the toenails or fingernails
* Any of the following in the 4 weeks (or as indicated) prior to randomization:
* Major surgery for any indication
* Any personal history of:
* Invasive cancer diagnosed or treated within the past 5 years. Participants who have been in remission for 5 years or more and have not required treatment in the past 5 years may be eligible if the principal investigator believes there is little to no risk of recurrence.
* Concurrent use of the following medications or treatments
* Other topical antifungals for any concomitant infection
* Females who are pregnant or lactating. Should a woman become pregnant or suspect she is pregnant while she is participating in this study she should notify the study physician immediately.
* Uncontrolled concurrent illness including ongoing or active infection, psychiatric illness or social situations that would limit compliance with study requirements or other underlying serious medical condition which, in the investigator's opinion, might preclude study participation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each patient served as their own control. One big toenail received nail polish only and the other big toenail was treated with nail polish and efinaconazole solution.
Units Other Than Participants: great toenail
Groups:
- Efinaconazole Solution and Nail Polish: Efinaconazole Solution and Nail Polish only (no base coat and no top coat) applied to great toenail
- Nail Polish Only: No efinaconazole applied to one great toe. Only Nail per treatment arm
- Efinaconazole Solution, Nail Polish, Top Coat, and Base Coat: One big toe will receive application of Efinaconazole solution on top of nail polish with base coat and top coat.
Period: Overall Study
Arm/Group | Efinaconazole Solution and Nail Polish | Nail Polish Only | Efinaconazole Solution, Nail Polish, Top Coat, and Base Coat | Nail Polish + Top Coat + Efinaconazole Solution
Started | 5; 5 great toenail | 5; 5 great toenail | 5; 5 great toenail | 5; 5 great toenail
Nail Polish | 5; 5 great toenail | 5; 5 great toenail | 5; 5 great toenail | 5; 5 great toenail
Nail Polish, Base Coat | 5; 5 great toenail | 5; 5 great toenail | 5; 5 great toenail | 5; 5 great toenail
Nail Polish, Top Coat | 5; 5 great toenail | 5; 5 great toenail | 5; 5 great toenail | 5; 5 great toenail
Completed | 5; 5 great toenail | 5; 5 great toenail | 5; 5 great toenail | 5; 5 great toenail
Not Completed | 0; 0 great toenail | 0; 0 great toenail | 0; 0 great toenail | 0; 0 great toenail

BASELINE CHARACTERISTICS:
Population: Healthy adult with large toenail present
Groups:
- Jublia: Both big toes will receive application of toenail polish. One big toe will not use Jublia.
  Jublia: Application of Jublia to one big toenail
  Nail polish: Application of nail polish to both big toe nails
  Subjects had to be healthy and have a big toenail
Arm/Group | Jublia
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Observe Stability of Nail Polish as Evidenced by Serial Photography With Efinaconazole Application in Terms of Days
Description: Observation: Serial photographs were combined with patient reported outcomes to assess the stability of self-applied toenail polish when efinaconazole was applied topically to the nail. (Expected stability of polish less than 14 days with application of Jublia as compared to nails without Jublia application)
Time Frame: Baseline to 14 days
Population: Healthy adults with normal appearing big toenails applied toenail polish to both big toes. Jublia was applied to one big toe daily on top of the nail polish. Serial photography and participant report demonstrated the day until the nail polish degraded (became damaged). Control results were not analyzed.
Measure: Median (Standard Deviation); unit: days of stability
Units Other Than Participants: nail polish cycle
Groups:
- Nail Polish and Efinaconazole Solution: Nail polish and Efinaconazole solution application (daily application of Efinaconazole solution)
- Efinaconazole Solution, Nail Polish, and Top Coat: Efinaconazole solution applied daily to nail with top coat and nail polish
- Placebo Comparator: Nail Polish Only: Both big toes will use nail polish only
- Base Coat + Nail Polish + Top Coat + Efinaconazole Solution: Active Comparator: Base Coat + Nail Polish + Top Coat + Efinaconazole Solution One big toe will receive application of Efinaconazole solution on top of nail polish with base coat and top coat.
Arm/Group | Nail Polish and Efinaconazole Solution | Efinaconazole Solution, Nail Polish, and Top Coat | Placebo Comparator: Nail Polish Only | Base Coat + Nail Polish + Top Coat + Efinaconazole Solution
Number analyzed (Participants) | 5 | 5 | 5 | 5
Number analyzed (nail polish cycle) | 15 | 15 | 15 | 15
days of stability | 1.5 (0.5) | 5 (2) | 15 (0) | 5 (2)

ADVERSE EVENTS:
Time Frame: 50 nail application cycles, 14 days of jublia application.
Groups:
- Jublia: Both big toes will receive application of nail polish. . Only one big toe will use efinaconazole.
  Jublia: Application of Jublia to one big toes
  Nail polish: Application of nail polish to both big toe nails
  Subjects had to be healthy and have a big toenail
Arm/Group | Jublia
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03022916/Prot_SAP_000.pdf